CLINICAL TRIAL: NCT00877773
Title: Histology-Independent Study of the mTOR Inhibitor, Temsirolimus, in Patients With Advanced Cancer
Brief Title: Phosphatidylinositol 3 Kinase and Mammalian Target of Rapamycin (PI3K-mTOR) in Advanced Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0827; NCI-2012-01265 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Cancers
Keywords: Advanced cancer; Advanced Cancer with genetic mutation; Phosphoinositides 3-kinase; PI3K; PIK3 mutations; Temsirolimus; CCI-779; Torisel; mTOR inhibitor
MeSH Terms: interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (Experimental): Temsirolimus 25 mg by vein over 60 minutes on Days 1, 8, 15, and 22 of each 4-week study cycle.
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — 25 mg by vein over 60 minutes on Days 1, 8, 15, and 22 of each 4-week study cycle.
  Other Names: CCI-779; Torisel

SUMMARY:
The goal of this clinical research study is to learn if temsirolimus can help to control advanced cancer in patients who also have a PI3K mutation and/or PTEN loss. The safety of this drug will also be tested.

DETAILED DESCRIPTION:
The Study Drug:

Temsirolimus is designed to block the growth of cancer cells, which may cause the cancer cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive temsirolimus through a needle in your vein on Days 1, 8, 15, and 22 of each 4-week study cycle. On Day 1 of Cycle 1, the study drug will be given over 60 minutes. If you tolerate the study drug well on Day 1 of Cycle 1, it will be given over 30 minutes at all other scheduled administration dates as long as you still tolerate it well. If the dose is not well tolerated, the dose will be reduced for future study visits.

You will receive Benadryl (diphenhydramine) or a similar drug by vein to help prevent side effects about 30 minutes before you receive the study drug.

Study Visits:

One (1) time each week (on each day that the study drug is being given), the following tests and procedures will be performed:

* Your weight and vital signs will be measured.
* You will be asked about any drugs you may be taking and about any side effects you may be having.
* Blood (about 2 teaspoons each time) will be drawn for pharmacodynamic (PD) testing. PD testing measures how the level of study drug in your body may affect the disease. This blood will be drawn at the following times:

At 8 hours (+/- 3 hours) after the dose At 24 hours (+/- 3 hours) after the dose At 72 hours (+/- 24 hours) after the dose

Every 2 weeks, blood (about 2 teaspoons) will be drawn for routine tests.

Every 4 weeks, you will have a physical exam; women who are able to become pregnant will also have a blood (about 1 teaspoon) pregnancy test.

Every 8 weeks, you will have a CT scan, MRI scan, and/or PET/CT scan to check the status of the disease.

Length of Study:

You will be on study for as long as you are benefiting or the disease is stable. You will be taken off study if the disease gets worse, you have intolerable side effects, or the study doctor thinks it is in your best interest.

End-of-Study Visit:

After you have finished taking the study drug, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and about any side effects you may be having.

This is an investigational study. Temsirolimus is FDA-approved and commercially available for the treatment of advanced renal cancer. Its use in other types of cancer is investigational.

Up to 65 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or has no standard therapy that improves survival by at least 3 months (unless temsirolimus is indicated as standard treatment for that disease).
2. Patients must have evaluable tumor(s) with documented PIK3 mutation and/or PTEN loss.
3. Patients must have creatinine </= 3 X upper limit of normal (ULN); absolute neutrophil count >/= 1,000/mL; platelets >/= 50,000; bilirubin </= 3.0 gm/dL. Except for patients with liver metastases: total bilirubin </= 5 ULN.
4. Women of childbearing potential must have a negative baseline blood pregnancy test. Women and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study.
5. Patients must be off other anti-tumor agents for at least 5 half lives of the agent or 4 wks from the last day of treatment, whichever is shorter. For cytotoxic therapies, patients should be off treatment for 3 or more weeks.
6. Patients may not be receiving any other experimental agents that are not FDA approved.
7. Ability to understand and willingness to sign a written consent document.
8. Treatment on this study may begin within 24 hours after Phase 0 dose of Temsirolimus.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with creatinine clearance <10 mL/min
3. Patients with a known hypersensitivity to any of the components or metabolites of the drug products.
4. Patients with major surgery within 30 days prior to entering study.
5. Patients on inhibitors or inducers of CYP3A4 metabolism will have the inhibitors or inducers stopped unless clinically contraindicated. See section 6 (Concomitant Medications) and Appendix E of the protocol for details.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Karp, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 6, 2009 to March 28, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Temsirolimus
Started | 44
Completed | 0 (No participant reached to first restaging.)
Not Completed | 44
Not completed — Disease Progression | 44

BASELINE CHARACTERISTICS:
Arm/Group | Temsirolimus
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 57 [16 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: For solid tumors, initial responses defined by Response Evaluation Criteria in Solid (RECIST) criteria in the evaluable lesion(s) per Complete Response (CR): Disappearance of all target lesions; confirmed at 4 weeks; Partial Response (PR): At least 30% decrease; confirmed at 4 weeks; Stable Disease (SD): Neither PR nor PD criteria met; Progressive Disease (PD): 20% increase; no CR, PR or SD documented before increased disease, or new lesion(s).
Time Frame: Baseline to Disease Progression (restaged at 8 weeks and at 4 months)
Population: Of the 44 participants enrolled, only 30 were evaluable for response.
Measure: Number; unit: participants
Arm/Group | Temsirolimus
Number analyzed (Participants) | 30
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 2
  Stable Disease | 20
  Progressive Disease (PD) | 8

ADVERSE EVENTS:
Time Frame: Adverse event collection through 2 cycles (about 8 weeks) of treatment.
Arm/Group | Temsirolimus
Serious Adverse Events (participants affected / at risk) | 6/44
Other Adverse Events (participants affected / at risk) | 19/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus (N=44)
Symptomatic Hydrocephalous (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncopal Episode (Nervous system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — with gram-negative rods
Cachexia (General disorders) | 1 (1)
Ventilatory Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus (N=44)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Neutropenia (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Hypotension (Cardiac disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Tongue Swelling (Gastrointestinal disorders) | 1 (1)
Acute Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Increased Swelling of the Face (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Partial Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Right-Sided Upper Extremity Weakness (General disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Increased Ascites (Gastrointestinal disorders) | 1 (1)
Syncopal Episode (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Unbalanced (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Brain Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fever (General disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Epitaxis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes